CLINICAL TRIAL: NCT06090877
Title: Role of Ultrasound and Shear Wave Elastography in Diagnosis and Grading of Cubital Tunnel Syndrome
Brief Title: US and Shear Wave Elastography in Cubital Tunnel Syndrome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eman Sayed Abdul Monem, dr, Assiut University
Other Study IDs: US in cubital tunnel syndrome
Record Dates: First submitted 2023-10-14; First posted 2023-10-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Ulnar Nerve Compression
Keywords: US+shear wave elstography+cubital tunnel syndrome
MeSH Terms: conditions — Ulnar Nerve Compression Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: US and shear wave elstography — using B mode US to assess ulnar nerve echogenicity, measuring its cross sectional area and assess any other anatomical abnormalites Measuring ulnar nerve stiffness using shear wave elastography All measurements done at the cubital tunnel, 2 cm proximal and distal to it compare findings with electrodiagnostic studies and intra operative findings
  Other Names: electrodiagnostic studies and suitable operation

SUMMARY:
This study aims to assess the role of US and SWE in diagnosis of CuTS and localization of its underlying etiology and verifying whether it can be diagnosed and graded based on US findings, especially quantitaive ulnar nerve stiffness data obtained using SWE, compared to ENMG and intraoperative findings (as gold standard)

DETAILED DESCRIPTION:
Ulnar nerve (UN) entrapment at the elbow is the second most frequent tunnel syndrome, following carpal tunnel syndrome.

Cubital tunnel syndrome (CuTS) is a common nerve entrapment syndrome of the upper extremity, caused by compression of the ulnar nerve at the cubital tunnel of the elbow.

The presentation of cubital tunnel syndrome varies, ranging from mild sensory symptoms to debilitating functional loss.

Typical CuTS symptoms include numbness, tingling, and dysesthesia in the ring, small finger and dorsum of the hand. As the disease progresses, atrophy of the hypothenar and first dorsal interosseous muscles occurs, which may interfere with daily activities. CuTS is likelier to be at an advanced stage at the time of intervention than carpal tunnel syndrome (CTS). Therefore, early diagnosis and treatment are important.

Also, due to anatomic variations, a broad spectrum of differential diagnosis, and miscellaneous clinical presentations, the clinical diagnosis is often far from straightforward. If not treated timely and adequately, CuTS can progress to persistent impairment of sensation, paresis, and joint contracture.

This condition is typically diagnosed using patient's history, physical examination, and electrodiagnostic studies. However, because CuTS has a variety of clinical characteristics, it is difficult to differentiate it from other diseases that can affect the elbow joint based on clinical presentation and an electrodiagnostic study.

Electroneuromyography (ENMG) is the gold standard examination in CuTS, but sheds no light on etiology.

Although an electrodiagnostic study is considered the most important diagnostic test for CuTS, it has some critical drawbacks. It is time-consuming, causing pain and injury to patients due to needle insertion and electrical stimulation, provides limited information regarding lesion localization and structural abnormalities, and carries a strong possibility of false negative results.

Thus, complementary imaging studies such as magnetic resonance or high resolution ultrasound (HRU) imaging are required for the diagnosis of various neuropathies. Ultrasound imaging in particular supports the diagnosis of neuropathy by providing superior spatial resolution of small peripheral nerves, allowing for dynamic evaluation and detailed information regarding lesion localization in addition to advantages of being fast, cheap, non invasive and painless procedure.

Moreover, as a recently-developed ultrasound imaging technology, shear-wave elastography (SWE) has the potential to provide quantitative values for the soft tissue stiffness of tissues, including the muscle, tendon, joint capsule, benign soft tissue mass, and nerves, and to improve the diagnostic performance of ultrasound imaging for various nerve neuropathies.

SWE is also an advanced quantitative ultrasound technique that can be used to evaluate soft tissue elasticity. In compressive neuropathy, a higher pressure within the canal could cause ischemia, edema, inflammation, and finally fibrosis in the intraneural space and the synovium. All of these changes to the compressed nerve may result in increased nerve stiffness. Therefore, SWE could be a valuable complement in the diagnosis of compressive neuropathy.

So, SWE seems to be a new, reliable, and simple quantitative diagnostic technique to aid in the precise diagnosis of ulnar neuropathy at the cubital tunnel, and HRU proved to be an effective diagnostic tool for CuTS and its etiologies

ELIGIBILITY:
Inclusion Criteria:

* In this study patients referred from the orthopedic clinic with a clinical diagnosis of clinical cubital tunnel syndrome and having electrodiagnostic studies will be included

Exclusion Criteria:

* Lack of electrodiagnostic studies.
* Refuse to do surgery when indicated

Ages: 10 Years to 75 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patient preparation:
  • No specific preparations needed. 2. Study instruments:- All patients will undergo B-mode ultrasound and SWE using GE Logiq S8 ultrasound machine with 9L-D Linear Array Transducer, at the Radiology Department of Assiut University Hospital, Assuit University.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
US and shear wave elastography findings in diagnosis and grading of cubital tunnel syndrome | base line
  measuring cross sectional area and nerve stiffness of the ulnar nerve at cubital tunnel and 2 cm proximal and distal to it as well detection of any anatomical abnormalities, assessing ulnar nerve instability Then findings of US and shear wave elastography will be compared with clinical, electrodiagnostic studies results and intra oprative findings.

SECONDARY OUTCOMES:
diagnosis and grading of cubital tunnel syndrome | base line
  using electrodiagnostic studies as reference to reach cut off values for ulnar nerve cross sectional area and nerve stiffness

REFERENCES:
- [Background] Shinohara I, Inui A, Mifune Y, Nishimoto H, Yamaura K, Mukohara S, Yoshikawa T, Kato T, Furukawa T, Hoshino Y, Matsushita T, Kuroda R. Diagnosis of Cubital Tunnel Syndrome Using Deep Learning on Ultrasonographic Images. Diagnostics (Basel). 2022 Mar 4;12(3):632. doi: 10.3390/diagnostics12030632. PMID 35328185
- [Background] Power HA, Peters BR, Patterson JMM, Padovano WM, Mackinnon SE. Classifying the Severity of Cubital Tunnel Syndrome: A Preoperative Grading System Incorporating Electrodiagnostic Parameters. Plast Reconstr Surg. 2022 Jul 1;150(1):115e-126e. doi: 10.1097/PRS.0000000000009255. Epub 2022 May 10. PMID 35544306
- [Background] Mezian K, Jacisko J, Kaiser R, Machac S, Steyerova P, Sobotova K, Angerova Y, Nanka O. Ulnar Neuropathy at the Elbow: From Ultrasound Scanning to Treatment. Front Neurol. 2021 May 14;12:661441. doi: 10.3389/fneur.2021.661441. eCollection 2021. PMID 34054704
- [Background] Kim S, Lee GY. Evaluation of the ulnar nerve with shear-wave elastography: a potential sonographic method for the diagnosis of ulnar neuropathy. Ultrasonography. 2021 Jul;40(3):349-356. doi: 10.14366/usg.20101. Epub 2020 Aug 23. PMID 33115185
- [Background] Rempel DM, Diao E. Entrapment neuropathies: pathophysiology and pathogenesis. J Electromyogr Kinesiol. 2004 Feb;14(1):71-5. doi: 10.1016/j.jelekin.2003.09.009. PMID 14759752
- [Background] Qing C, Zhang J, Wu S, Ling Z, Wang S, Li H, Li H. Clinical classification and treatment of cubital tunnel syndrome. Exp Ther Med. 2014 Nov;8(5):1365-1370. doi: 10.3892/etm.2014.1983. Epub 2014 Sep 22. PMID 25289024